CLINICAL TRIAL: NCT06066502
Title: PREcision VENTilation to Attenuate Ventilator-Induced Lung Injury: A Phase 3 Multicenter Randomized Clinical Trial
Brief Title: Precision Ventilation vs Standard Care for Acute Respiratory Distress Syndrome
Acronym: PREVENT VILI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: NYU Langone Health (Other); Massachusetts General Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Daniel Talmor, Professor and Chair of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023P000682; 1U24HL166784 (NIH); 1UG3HL166785 (NIH)
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Acute Respiratory Distress Syndrome; Respiratory Failure
Keywords: critical care; critical illness; esophageal manometry; transpulmonary pressure; mechanical ventilation; lung stress
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency; Critical Illness

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the intervention arm or control arm.
  Participants in the intervention group (precision ventilation), will have mechanical ventilation using settings directed by the amount of air pressure in the chest and lungs, using esophageal manometry. The treating clinical team is not masked to esophageal and transpulmonary pressure values and can view these data throughout the period of protocol-directed ventilation.
  Participants in the control group (guided usual care), will have ventilator support (low tidal volume mechanical ventilation) managed by the clinical team per usual care. The treating clinical team is masked to esophageal and transpulmonary pressure values and cannot view or be informed of these data at any time during the period of protocol-directed ventilation. An esophageal catheter will be inserted strictly for monitoring of respiratory mechanics by study staff, but values will not be used to titrate the ventilator.
Who Masked: Participant
Masking Description: Study team and leadership will be blinded to all analyses throughout the study. Unblinded statistician will perform analyses for the Data and Safety Monitoring Board (DSMB) and be sequestered from the remainder of the team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Precision ventilation (Experimental): Ventilator support will be calibrated to maintain the range of lung stress typical of relaxed breathing in healthy adults. The ventilator management protocol takes into account pleural pressure, tidal volume and driving pressure, fraction of inspired oxygen (FiO2) and oxygen saturation (SpO2), and positive end-expiratory pressure (PEEP) titration.
  Interventions: Other: Precision ventilation
- Guided usual care (Active Comparator): Ventilator support will be managed by the clinical team per usual care with select protocol-based guard rails to avoid practice extremes beyond the current body of evidence. PEEP titration will be performed by the clinical team within the limits set in. The allowable combinations of PEEP and FiO2 in the control arm reflect pre-intervention usual care observed at baseline in the recent large federally-funded multicenter ARDS trials.
  Interventions: Other: Guided usual care ventilation

INTERVENTIONS:
Other: Precision ventilation — The intervention arm prioritizes mitigation of ventilator-induced-lung-injury by individualizing support to patient-specific mechanics in an integrated approach to limit overdistension and atelectrauma. This is accomplished in this arm by titration of tidal volume to limitation of driving pressure at 12 centimeters of water (cmH2O) or less and using esophageal manometry to titrate PEEP to a transpulmonary pressure of 0 cmH2O with adjustments in respiratory rate to allow for permissive hypercapnia and FiO2 adjustments to assure adequate oxygenation.
  Arms: Precision ventilation
Other: Guided usual care ventilation — The comparison arm allows clinician discretion when titrating PEEP and tidal volume, while setting general targets for allowable PEEP/FiO2 combinations, target range for SpO2, and target range for tidal volume. This arm applies routine best-practice guidelines. This includes maintenance of tidal volumes of 6-8 cc/kg of ideal body weight, limiting plateau pressures to 30 cmH2O or less and application of PEEP-FiO2 combinations which include a wide range of typical usual care with esophageal manometry only for data collection and not clinical adjustment.
  Arms: Guided usual care

SUMMARY:
The goal of this interventional study is to compare standard mechanical ventilation to a lung-stress oriented ventilation strategy in patients with Acute Respiratory Distress Syndrome (ARDS). Participants will be ventilated according to one of two different strategies. The main question the study hopes to answer is whether the personalized ventilation strategy helps improve survival.

DETAILED DESCRIPTION:
ARDS is a devastating condition that places a heavy burden on public health resources. Recent changes in the practice of mechanical ventilation have improved survival in ARDS, but mortality remains unacceptably high.

This application is for support of a phase III multi-centered, randomized controlled trial of mechanical ventilation, directed by driving pressure and esophageal manometry, in patients with moderate or severe ARDS. The primary hypothesis is that precise ventilator titration to maintain lung stress within 0-12 centimeters of water (cm H2O), the normal physiological range experienced during relaxed breathing, will improve 60-day mortality, compared to guided usual care.

Specific Aim 1: To determine the effect on mortality of the precision ventilation strategy, compared to guided usual care, in patients with moderate or severe ARDS.

• Hypothesis 1: The precision ventilation strategy will decrease 60-day mortality (primary trial endpoint).

Specific Aim 2: To evaluate the effects on lung injury of the precision ventilation strategy, compared to guided usual care, in patients with moderate or severe ARDS.

* Hypothesis 2a: The precision ventilation strategy will improve clinical pulmonary recovery, defined using the composite endpoint alive and ventilator-free (AVF).
* Hypothesis 2b: The precision ventilation strategy will attenuate alveolar epithelial injury.

Specific Aim 3: To evaluate the hemodynamic safety profile of the precision ventilation strategy, compared to guided usual care, in patients with moderate or severe ARDS.

• Hypothesis 3: The precision ventilation strategy will decrease hemodynamic instability, measured as shock-free days through Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Moderate or severe ARDS, defined as meeting all of the following (a-e):

   1. Invasive ventilation with positive end-expiratory pressure (PEEP) ≥ 5 cm H2O
   2. Hypoxemia as characterized by: • If arterial blood gas (ABG) available: the partial pressure of oxygen in the arterial blood (PaO2)/FiO2 ≤ 200 mm Hg, or, • if ABG not available OR overt clinical deterioration in oxygenation since last ABG: SpO2/FiO2 ≤ 235 with SpO2 ≤ 97% (both conditions) on two representative assessments between 1 to 6 hours apart. • If patient is positioned prone or receiving inhaled pulmonary vasodilator at time of screening:

      Qualifying PaO2/FiO2 or SpO2/FiO2 (as defined above) that was recorded within the 6 hours immediately prior to initiating either of these therapies may be used for eligibility determination. • If PEEP has been increased by > 5 cm H2O within the last 12 hours immediately prior to screening:

      Qualifying PaO2/FiO2 or SpO2/FiO2 (as defined above) prior to PEEP increase may be used for eligibility determination if recorded within this 12-hour window.
   3. Bilateral lung opacities on chest imaging not fully explained by effusions, lobar collapse, or nodules
   4. Respiratory failure not fully explained by heart failure or fluid overload
   5. Onset within 1 week of clinical insult or new/worsening symptoms
3. Early in ARDS course

   * Full criteria for moderate-severe ARDS (#2 above) first met within previous 3 days
   * Current invasive ventilation episode not more than 4 days duration
   * Current severe hypoxemic episode (receipt of invasive ventilation, noninvasive ventilation, or high-flow nasal cannula) not more than 10 days duration

Exclusion Criteria:

1. Esophageal manometry already in use clinically
2. Severe brain injury: including suspected elevated intracranial pressure, cerebral edema, or Glasgow coma score (GCS) ≤ 8 directly caused by severe brain injury (e.g., ischemia or hemorrhage)
3. Gross barotrauma or chest tube inserted to treat barotrauma (note: chest tube inserted strictly for drainage of pleural effusion is not an exclusion)
4. Esophageal varix or stricture that, in judgement of the site investigator, significantly increases risk of esophageal catheter placement; recent oropharyngeal or gastroesophageal surgery; or past esophagectomy
5. Ongoing severe coagulopathy (platelet < 5000/μL or INR > 4)
6. Extracorporeal membrane oxygenation (ECMO) or CO2 removal (ECCO2R)
7. Neuromuscular disease that impairs spontaneous breathing (including but not limited to amyotrophic lateral sclerosis, Guillain-Barré syndrome, spinal cord injury at C5 or above)
8. Any of the following severe chronic lung diseases: continuous home supplemental oxygen > 3 liters/minute, pulmonary fibrosis, cystic fibrosis, lung transplant, or acute exacerbation of a chronic interstitial lung disease (ILD)
9. Severe shock: norepinephrine-equivalent dose ≥ 0.6 μg/kg/min or simultaneous receipt of ≥ 3 vasopressors
10. Severe liver disease, defined as Child-Pugh Class C (Section 12.3)
11. ICU admission for burn injury
12. Current ICU stay > 2 weeks or acute care hospital stay > 4 weeks
13. Estimated mortality > 50% over 6 months due to underlying chronic medical condition (e.g. metastatic pancreatic cancer) as assessed by the study physician
14. Moribund patient not expected to survive 24 hours as assessed by the study physician; if cardiopulmonary resuscitation (CPR) was provided, assessment for moribund status must occur at least 6 hours after CPR was completed
15. Current limitation on life-sustaining care (other than do-not-resuscitate), or expectation by clinical team that a limitation on life-sustained care will be adopted within next 24 hours.
16. Treating clinician refusal or unwilling to use protocol-specified ventilator settings/modes
17. Prisoner
18. Previous enrollment in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
60-day mortality | 60 days from trial enrollment
  All-cause, all-location mortality

SECONDARY OUTCOMES:
28-day mortality | 28 days from trial enrollment
  All-cause, all-location mortality
Alive and ventilator-free through 28 days | 28 days from trial enrollment
  A composite outcome that incorporates survival for the defined follow-up interval and time to successful liberation from invasive mechanical ventilation (IMV) among survivors.
Alive and Respiratory Support-Free | 28 days from trial enrollment
  A composite outcome that incorporates survival for the defined follow-up interval and time to successful liberation from advanced respiratory support among survivors. Advanced respiratory support is defined in Section 1.2. This outcome will be formulated as a win ratio and separately as a time-to-event competing risk endpoint.
Barotrauma through Day 14 | 14 days from trial enrollment
  Any occurrence of pneumothorax, pneumomediastinum, subcutaneous emphysema, or chest tube insertion for barotrauma through Day 14 or until successful liberation from IMV, whichever occurs first.

OTHER OUTCOMES:
Hemodynamic Instability Index through Hour 4 and daily through Day 7 | From hour 4 through Day 7 from enrollment
  A hemodynamic instability index will be computed per a six-level ordinal scale
Shock-free days through Day 28 | 28 days from trial enrollment
  The number of days, regardless of consecutiveness, during which vasopressors have not been administered for at least 1 uninterrupted hour, through Day 28.
Duration of vasopressor support through Day 28 | 28 days from trial enrollment
  A component of the shock-free days composite outcome, calculated as number of days, regardless of consecutiveness, during which the patient required vasopressor support for at least 1 uninterrupted hour of the day.
Renal failure-free days through Day 28 | 28 days from trial enrollment
  The number of days between successful liberation from renal replacement therapy and Day 28.
Refractory hypoxemia through Day 14 | 14 days from trial enrollment
  Any occurrence of SpO2 < 88% continuously for at least 30 minutes' duration despite valid pulse-oximetry waveform and protocol-directed ventilatory support, through Day 28 or until successful liberation from IMV, whichever occurs first.
Refractory acidemia through Day 14 | 14 days from trial enrollment
  Any occurrence of arterial pH < 7.15 on two consecutive measures at least 30 minutes apart despite protocol-directed ventilatory support, through Day 28 or until successful liberation from IMV, whichever occurs first.
Daily Sequential Organ Failure Assessment (SOFA) through Day 7 | 7 days from trial enrollment
  SOFA will be computed daily for live patients through Day 7, omitting Glasgow Coma Scale element.
ICU length of stay | 60 days
  Number of days in the ICU from enrollment until the last transfer out of ICU, hospital discharge, death, or Day 60, whichever occurs first. The "last day" method will be used: if a participant leaves the ICU but is then transferred back into the ICU during the same hospitalization within the 60-day follow up period, the brief time interval outside the ICU will count toward ICU length of stay.
Hospital length of stay | 60 days
  Number of days in the hospital from enrollment until hospital discharge, death, or Day 60, whichever occurs first.
Alveolar epithelial injury biomarkers | 2 days from trial enrollment
  The change in plasma levels of Plasma Soluble Receptor for Advanced glycation end-products (sRAGE) and surfactant protein D (SP-D) will be compared between baseline and Day 2.
Pro-fibrosis biomarkers | 2 days from trial enrollment
  The change in plasma levels of Plasma procollagen-III N-terminal peptide (P3NP) and matrix metalloproteinase-7 (MMP7) will be compared between baseline and Day 2.
Endothelial barrier function biomarkers | 2 days from trial enrollment
  The change in plasma levels of Plasma angiopoietin-2 and vascular endothelial growth factor receptor 1 (VEGFR1, also known as FLT1) will be compared between baseline and Day 2.
Inflammatory biomarkers | 2 days from trial enrollment
  The change in plasma levels of Plasma interleukin-6 (IL6) and interleukin-8 (IL8) will be compared between baseline and Day 2.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Talmor, MD MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (24):
- United States (24):
  - University of Arizona, Tucson, Arizona
  - University of California, San Diego, La Jolla, California
  - University of California, Los Angeles Medical Center, Los Angeles, California
  - Cedar-Sinai Medical Center, Los Angeles, California
  - University of California, San Francisco, San Franciso, California
  - University of Chicago, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - NYU Lagone Health, New York, New York
  - New York City Health + Hospitals/ Bellevue, New York, New York
  - Albert Einstein College of Medicine/Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Baylor College of Medicine / St. Luke's Medical Center, Houston, Texas
  - Intermountain Health, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - University of Washingont/Harborview Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Data will be made publicly available via the NHLBI Biologic Specimen and Data Repository Information Coordinating Center (BioLINCC) repository. As per BioLINCC policy, data will be submitted within one year of completion of the final follow up assessment, or within one year of primary manuscript publication, whichever comes first.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available within one year of completion of the final follow up assessment, or within one year of primary manuscript publication, whichever comes first. Data will be available for 10 years.
Access Criteria: Outside investigators who wish to use data will submit a formal request, including rationale, analysis plan, and local Institutional Review Board (IRB) determination. The PREVENT VILI Executive Committee will review and respond to all requests. All data sharing will be codified by the appropriate contract / data use agreement. Recipient researchers must promise in writing to never attempt to access identifiable health/medical information or to attempt to identify the subject(s) who provided the specimen/data. Any intent to use materials or data for commercial purposes must be clearly disclosed as part of the request.

REFERENCES:
- [Background] Beitler JR, Sarge T, Banner-Goodspeed VM, Gong MN, Cook D, Novack V, Loring SH, Talmor D; EPVent-2 Study Group. Effect of Titrating Positive End-Expiratory Pressure (PEEP) With an Esophageal Pressure-Guided Strategy vs an Empirical High PEEP-Fio2 Strategy on Death and Days Free From Mechanical Ventilation Among Patients With Acute Respiratory Distress Syndrome: A Randomized Clinical Trial. JAMA. 2019 Mar 5;321(9):846-857. doi: 10.1001/jama.2019.0555. PMID 30776290
- [Background] National Heart, Lung, and Blood Institute PETAL Clinical Trials Network; Moss M, Huang DT, Brower RG, Ferguson ND, Ginde AA, Gong MN, Grissom CK, Gundel S, Hayden D, Hite RD, Hou PC, Hough CL, Iwashyna TJ, Khan A, Liu KD, Talmor D, Thompson BT, Ulysse CA, Yealy DM, Angus DC. Early Neuromuscular Blockade in the Acute Respiratory Distress Syndrome. N Engl J Med. 2019 May 23;380(21):1997-2008. doi: 10.1056/NEJMoa1901686. Epub 2019 May 19. PMID 31112383